CLINICAL TRIAL: NCT06485232
Title: An Exploratory Study on the Safety and Efficacy of Universal CAR-T Cells Targeting BCMA and CD19 in the Treatment of Refractory Autoimmune Diseases of the Nervous System
Brief Title: Universal CAR-T Cells in Patients with Refractory Autoimmune Diseases of the Nervous System.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Bioray Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-BRL-302-02
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Myasthenia Gravis, Generalized; Multiple Sclerosis; Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: universal CAR-T; Neuromyelitis Optica Spectrum Disorders; Myasthenia Gravis; Multiple Sclerosis; Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Neuromyelitis Optica; Myasthenia Gravis; Multiple Sclerosis; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BCMA CAR-T Group (Experimental): Universal BCMA CAR-T
  Interventions: Drug: Universal BCMA CAR-T
- CD19 CAR-T Group (Experimental): Universal CD19 CAR-T
  Interventions: Drug: Universal CD19 CAR-T
- BCMA CAR-T + CD19 CAR-T Group (Experimental): Universal BCMA CAR-T; Universal CD19 CAR-T
  Interventions: Drug: Universal BCMA CAR-T; Universal CD19 CAR-T

INTERVENTIONS:
Drug: Universal BCMA CAR-T — Universal BCMA CAR-T
  Arms: BCMA CAR-T Group
Drug: Universal CD19 CAR-T — Universal CD19 CAR-T
  Arms: CD19 CAR-T Group
Drug: Universal BCMA CAR-T; Universal CD19 CAR-T — Universal BCMA CAR-T; Universal CD19 CAR-T
  Arms: BCMA CAR-T + CD19 CAR-T Group

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 25 participants with refractory autoimmune diseases of nervous system. This study aims to evaluate the safety and efficacy of the treatment with universal BCMA and CD19 CART.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years (for MS patients, 18-55 years); both genders eligible.
* Subjects with refractory neurological autoimmune diseases who have failed standard treatment or lack effective treatment, Including neuromyelitis optica spectrum disorders(NMOSD), generalized myasthenia gravis(gMG), chronic inflammatory demyelinating Polyradiculoneuropathy(CIDP) and multiple sclerosis(MS).
* Anticipated survival of ≥ 12 weeks as judged by the researcher.
* Agrees to use double barrier methods, condoms, oral or injectable contraceptives, or intrauterine devices during the study period and for one year after taking the study medication.
* Provides written informed consent.

Exclusion Criteria:

* History of solid organ transplantation.
* Malignant tumor within the last two years.
* Positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb), with peripheral blood Hepatitis B virus (HBV) DNA detected as positive; positive for Hepatitis C virus antibodies, with peripheral blood Hepatitis C virus RNA detected as positive; positive for Human Immunodeficiency Virus (HIV) antibodies; positive for Cytomegalovirus (CMV) DNA; positive for syphilis.
* Primary immunodeficiency (congenital or acquired).
* Severe cardiac disease.
* History of psychiatric disorders or history of psychotropic drug abuse, with no history of withdrawal.
* Allergic constitution or a history of severe allergies.
* Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities(DLTs) | First 28 days after infusion
  Incidence of dose-limiting toxicities(DLTs)
Incidence of adverse events(AEs) and severe adverse | Up to 12 months after infusion
  Incidence of adverse events(AEs) and severe adverse events(SAEs).

SECONDARY OUTCOMES:
Concentrations of UCAR-T cells | 3 months
  The concentration of BCMA UCAR T cells and CD19 UCAR-T cells in peripheral blood after infusion
B cell levels in peripheral blood | 3 months
  The change of B cell levels in peripheral blood after infusion
Changes of pathogenic antibody titers after infusion | 1, 3, 6 ,12months
  The changes of pathogenic antibody titers in peripheral blood or cerebrospinal fluid.
NMOSD: Annualized relapse rate | 6, 12months
  ARR is defined as the number of relapses divided by the total participant-years after infusion
gMG: Changes of Myasthenia Gravis Activities if Daily Living (MG-ADL) Score | 1, 3, 6, 12months
  MG-ADL scale assesses the impact of gMG on daily functions by measuring 8 signs or symptoms that are commonly affected in gMG. Each item is measured on a 4-point scale, where a score of 0 represents normal function and a score of 3 represents the loss of ability to perform that function. Total scores range from 0 to 24 points, with a higher score showing more severe gMG.
CIDP:Changes of Inflammatory Neuropathy Cause and Treatment (INCAT) Score after infusion. | 1, 3, 6, 12months
  The INCAT score assesses the functionality of the arms and legs by giving a 0-5 score for arms and legs, with 0 representing no disability and 5 representing no arm function or inability to stand/walk.
MS: Changes of the number of Gd-enhancing T1 Lesions | 6, 12months
  The changes of enhancing Lesions as detected by brain Magnetic Resonance Imaging (MRI)
MS: Changes of the number of Number of New or Enlarging T2 Lesions | 6, 12months
  Number of new/enlarging T2 lesions on last available MRI scan compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No